CLINICAL TRIAL: NCT00678249
Title: A Prospective, Multi-Center, Randomized Evaluation of an IMPRA/Bard ePTFE Encapsulated Carbon Lined Nitinol Endoluminal Device for AV Access Graft Stenoses
Brief Title: Pivotal Study for the FLAIR Endovascular Stent Graft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: John Reviere, Director, Clinical Affairs, Bard Peripheral Vascular, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMP-9809; P060002 (Other: Food and Drug Administration)
Record Dates: First submitted 2008-05-13; First posted 2008-05-15 (Estimated); Results first posted 2011-05-09 (Estimated); Last update posted 2011-05-11 (Estimated); Status verified 2011-05

CONDITIONS: Stenoses
Keywords: Hemodialysis; Vascular Prosthesis; stenoses; grafts
MeSH Terms: conditions — Constriction, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- FLAIR (Experimental): Primary PTA followed by placement of the FLAIR Endovascular Stent Graft
  Interventions: Device: FLAIR Endovascular Stent Graft
- PTA Only (Active Comparator): Percutaneous Transluminal Angioplasty
  Interventions: Procedure: PTA
- FLAIR Roll-in Participants (Experimental): Primary Patency followed by placement of the FLAIR Endovascular Stent Graft. Roll-in participants were enrolled in the study for training purposes and were not randomized.
  Interventions: Device: FLAIR Endovascular Stent Graft

INTERVENTIONS:
Device: FLAIR Endovascular Stent Graft — Primary balloon angioplasty followed by placement of the FLAIR Endovascular Stent Graft
  Other Names: Flair; Stent Graft
  Arms: FLAIR
Procedure: PTA — Percutaneous Transluminal Angioplasty
  Other Names: Flair; Stent Graft
  Arms: PTA Only
Device: FLAIR Endovascular Stent Graft — Primary PTA followed by placement of the FLAIR Endovascular Stent Graft. Roll-in participants were enrolled in the study for training purposes and were not randomized.
  Other Names: Flair; Stent Graft
  Arms: FLAIR Roll-in Participants

SUMMARY:
This study compared the FLAIR™ Endovascular Stent Graft to balloon angioplasty in patients with stenoses at the venous anastomosis of a synthetic AV access graft.

DETAILED DESCRIPTION:
A total of 227 patients were treated at 16 U.S. investigational sites to evaluate the safety and effectiveness of the FLAIR™ Endovascular Stent Graft. This study compared the FLAIR™ Endovascular Stent Graft to balloon angioplasty in patients with stenoses at the venous anastomosis of a synthetic AV access graft.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients between 18 to 90 years of age whose hemodialysis access was a synthetic AV access graft located in an arm.
* Angiographic evidence of one or more stenoses, 7 cm or less in length and greater than or equal to 50%, at the graft-vein anastomosis of a synthetic AV access graft. The entire lesion must have been located within 7 cm of the anastomosis such that approximately 1 cm of the IMPRA/Bard Device must have extended into non-diseased vein and approximately 1 cm, but no more than 2 cm, of the IMPRA/Bard Device will be extended into non-diseased AV graft.
* Clinical evidence of a hemodynamically significant stenosis.
* Percutaneous endovascular therapy for the identified lesion was the best treatment choice in the opinion of the investigator.
* Patients must have been able to understand and provide informed consent.
* Patients whose synthetic AV access grafts had been implanted greater than 30 days and had undergone 1 or more successful hemodialysis sessions.
* During primary balloon angioplasty, full expansion of an appropriately sized angioplasty balloon, in the operator's judgment, must have been achieved.

Exclusion Criteria:

* Concomitant disease (e.g., terminal cancer) or other medical condition that was likely to result in death of the patient within 6 months of the time of implantation.
* Stenoses that had a corresponding thrombosis treated within 7 days.
* The presence of a second lesion in the access circuit less than or equal to 3 cm from the edges of the primary lesion that was treated within 30 days or that was greater than or equal to 30%. Access circuit was defined as the area from the AV access graft arterial anastomosis to the superior vena cava-right atrial junction.
* The presence of a second lesion in the access circuit greater than 3 cm from the edges of the primary lesion that was greater than or equal to 30%. Second lesions that were greater than or equal to 30% must have been treated prior to patient inclusion to reduce the percent stenosis to less than 30%.
* Patients who were unwilling or unable to return for follow-up visits or patients with whom follow-up visits may have been unreliable.
* Patients who had a stent placed at the target lesion site.
* Patients with a blood coagulative disorder or sepsis.
* Patients in which the IMPRA/Bard Device would have been required to cross an angle (between the inflow vein and synthetic AV access graft) that was greater than 90 degrees.
* Patients in which the IMPRA/Bard Device would have been required to be deployed fully across the elbow joint, which is identified radiographically by a combination of the humeroulnar joint and the humeroradial joint.
* Patients with a contraindication to the use of contrast media.
* Patients whose AV access graft was infected.
* Patients who were currently or were scheduled to enroll in other investigations that conflicted with follow-up testing or confounds data in this trial.
* Procedural use of another investigational device.
* Patients who were pregnant.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2001-01; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Ciavarella, MD, Study Director — C. R. Bard
Locations (1):
- New York Presbyterian Hospital/Columbia, New York, New York, United States

REFERENCES:
- [Derived] Haskal ZJ, Trerotola S, Dolmatch B, Schuman E, Altman S, Mietling S, Berman S, McLennan G, Trimmer C, Ross J, Vesely T. Stent graft versus balloon angioplasty for failing dialysis-access grafts. N Engl J Med. 2010 Feb 11;362(6):494-503. doi: 10.1056/NEJMoa0902045. PMID 20147715

RESULTS

PARTICIPANT FLOW:
Groups:
- FLAIR Roll-In Participants: Primary PTA followed by placement of the FLAIR Endovascular Stent Graft. Roll-in participants were enrolled in the study for training purposes and were not randomized.
Period: Overall Study
Arm/Group | FLAIR | PTA Only | FLAIR Roll-In Participants
Started | 97 | 93 | 37
Completed | 97 | 93 | 37
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FLAIR | PTA Only | FLAIR Roll-In Participants | Total
Number analyzed (Participants) | 97 | 93 | 37 | 227
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 52 | 50 | 21 | 123
  >=65 years | 45 | 43 | 16 | 104
Age Continuous [Mean (Standard Deviation); unit: years] | 61.83 (14.63) | 59.83 (13.58) | 62.16 (11.84) | 60.36 (14.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 57 | 23 | 144
  Male | 33 | 36 | 14 | 83
Region of Enrollment [Number; unit: participants]
  United States | 97 | 93 | 37 | 227

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Treatment Area Primary Patency (TAPP)
Description: TAPP was defined as patency (open to blood flow) after the study index procedure until reintervention in the treatment area (within 5 mm proximal or 5 mm distal to the study device or index balloon angioplasty treatment area), or thrombotic occlusion that involved the treatment area.
Time Frame: 6 month follow-up
Population: If a participant was lost to follow-up prior to the follow-up interval window, then the participant's status was considered missing for that time point and was not included in the ITT analysis.
Measure: Number; unit: Percentage of Participants
Arm/Group | FLAIR | PTA Only | FLAIR Roll-In Participants
Number analyzed (Participants) | 91 | 86 | 35
Percentage of Participants | 51 | 23 | 60
Statistical Analysis 1: Comparison: FLAIR vs PTA Only; Test type: Superiority or Other; p < 0.001, Regression, Logistic

2. Secondary Outcome: Total Number of Adverse Events
Description: The safety endpoint was evaluated based on the incidence of adverse events observed within the same time interval. An adverse event was defined as any undesirable clinical occurrence in a patient that (a) is considered possibly or definietly device related by the investigator, (b) involves the access circuit (AV graft arterial anastomosis to the superior vena cava-right atrial junction) or the arm where the access circuit is located or (c) the investigator considers relevant to the objectives of this study. An adverse event could be mild, moderate or severe.
Time Frame: 6 month Follow-Up
Measure: Number; unit: total events
Arm/Group | FLAIR | PTA Only | FLAIR Roll-In Participants
Number analyzed (Participants) | 97 | 93 | 37
total events | 106 | 106 | 33

3. Secondary Outcome: Percent of Participants With Successful Delivery of the Device
Description: The ability to successfully deliver the FLAIR™ Endovascular Stent Graft. Successful delivery is the ability to deliver and seat the implant in the intended location of a stenosed segment of the venous anastomosis region of a synthetic access graft. This attribute is only applicable to the FLAIR and FLAIR Roll-in arms.
Time Frame: Index Procedure
Population: The PTA Only group was not analyzed for this outcome measure because it is for successful delivery of the FLAIR study device (PTA Only is the control arm).
Measure: Number; unit: Percentage of Participants
Arm/Group | FLAIR | PTA Only | FLAIR Roll-In Participants
Number analyzed (Participants) | 97 | 0 | 37
Percentage of Participants | 99 |  | 100

4. Secondary Outcome: Percent of Participants With Procedural Success
Description: Procedural Success was defined as anatomic success (<30% residual stenosis) and at least one indicator of hemodynamic or clinical success
Time Frame: Index Procedure
Measure: Number; unit: Percentage of Participants
Arm/Group | FLAIR | PTA Only | FLAIR Roll-In Participants
Number analyzed (Participants) | 97 | 93 | 37
Percentage of Participants | 94 | 73 | 95

5. Secondary Outcome: Percent of Participants With TAPP
Description: as for outcome 1
Time Frame: 2 month Follow-Up
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | FLAIR | PTA Only | FLAIR Roll-In Participants
Number analyzed (Participants) | 96 | 92 | 37
Percentage of Participants | 80 | 77 | 89

6. Secondary Outcome: Percent of Participants With Access Circuit Primary Patency (ACPP)
Description: ACCP defined as patency (open to blood flow) following the index study procedure until access thrombosis or an intervention of a lesion anywhere within the access circuit.
Time Frame: 6 month Follow-Up
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | FLAIR | PTA Only | FLAIR Roll-In Participants
Number analyzed (Participants) | 92 | 86 | 35
Percentage of Participants | 38 | 20 | 43

7. Secondary Outcome: Percent of Participants With Access Circuit Assisted Primary Patency (ACAPP)
Description: ACAPP defined as patency (open to blood flow)following the index study procedure until access thrombosis or a surgical intervention that excludes the treated lesion from the access circuit.
Time Frame: 6 month Follow-Up
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | FLAIR | PTA Only | FLAIR Roll-In Participants
Number analyzed (Participants) | 90 | 84 | 35
Percentage of Participants | 66 | 74 | 66

8. Secondary Outcome: Percent of Participants With Access Circuit Cumulative Patency (ACCP or Secondary Patency)
Description: ACCP defined as patency (open to blood flow) following the index study procedure until the access is surgically revised or abandoned because of the inability to treat the original lesion. Multiple treatments for occlusions to restore patency are compatible with ACCP.
Time Frame: 6 month Follow-Up
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | FLAIR | PTA Only | FLAIR Roll-In Participants
Number analyzed (Participants) | 91 | 85 | 35
Percentage of Participants | 81 | 86 | 91

9. Secondary Outcome: Percent of Participants With Binary Restenosis
Description: Binary restenosis defined as lesions with greater than or equal to 50% diameter stenosis of the treatment area (calculated by a core lab).
Time Frame: 6 month Follow-Up
Population: If a participant was lost to follow-up prior to the follow-up interval window (or the core lab could not assess the angiogram), then the participant's status was considered missing for that time point and was not included in the ITT analysis.
Measure: Number; unit: Percentage of Participants
Arm/Group | FLAIR | PTA Only | FLAIR Roll-In Participants
Number analyzed (Participants) | 76 | 67 | 28
Percentage of Participants | 28 | 78 | 25

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | FLAIR | PTA Only | FLAIR Roll-In Participants
Serious Adverse Events (participants affected / at risk) | 5/97 | 5/93 | 1/37
Other Adverse Events (participants affected / at risk) | 67/97 | 80/93 | 26/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | FLAIR (N=97) | PTA Only (N=93) | FLAIR Roll-In Participants (N=37)
Death (Cardiac disorders) | 5/95 (5) | 5/90 (5) | 1/36 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | FLAIR (N=97) | PTA Only (N=93) | FLAIR Roll-In Participants (N=37)
Infection (Infections and infestations) | 6/95 (6) | 2/90 (2) | 0/36 (0)
Stenosis (Vascular disorders) | 38/95 (38) | 69/90 (69) | 15/36 (15)
Thrombotic Occlusion (Vascular disorders) | 31/95 (31) | 19/90 (19) | 12/36 (12)
Vessel rupture (Vascular disorders) | 3/95 (3) | 1/90 (1) | 0/36 (0)
Pseudoaneurysm (Vascular disorders) | 5/95 (5) | 2/90 (2) | 1/36 (1)
Hematoma (Vascular disorders) | 2/95 (2) | 0/90 (0) | 0/36 (0)
Signficant arm or hand edema (Blood and lymphatic system disorders) | 3/95 (3) | 2/90 (2) | 1/36 (1)
Steal syndrome (Vascular disorders) | 2/95 (2) | 1/90 (1) | 1/36 (1)
Congestive heart failure (Cardiac disorders) | 4/95 (4) | 2/90 (2) | 1/36 (1)
Cerebrovascular accident (Nervous system disorders) | 2/95 (2) | 3/90 (3) | 0/36 (0)
Device migration (Surgical and medical procedures) | 4/95 (4) | 0/90 (0) | 0/36 (0)
Permanent deformation of the Endoluminal Device (Surgical and medical procedures) | 1/95 (1) | 0/90 (0) | 1/36 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No